CLINICAL TRIAL: NCT03154801
Title: Early Detection and Paramedical Care of Sexual Difficulties in Nervous System Diseases: Example of Multiple Sclerosis and Brain Tumors
Brief Title: Early Detection and Paramedical Care of Sexual Difficulties in Nervous System Diseases: Example of Multiple Sclerosis and Brain Tumors (NEUROSEX)
Acronym: NEUROSEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P140709
Record Dates: First submitted 2017-05-09; First posted 2017-05-16 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Low Grade Glioma of Brain; Multiple Sclerosis; Sexual Dysfunctions
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paramedical care (Experimental): paramedical early detection of sexual dysfunction and sexual health counseling
  Interventions: Other: Paramedical care

INTERVENTIONS:
Other: Paramedical care — Paramedical early detection of sexual dysfunction and sexual health counseling

SUMMARY:
This study aim to ensure that the implementation of a paramedical screening program and counseling in sexual health of patients with neurological pathologies (low-grade gliomas and Multiple Sclerosis) improves their sexual health.

ELIGIBILITY:
Inclusion Criteria:

1. Any major patient, followed in the GHPSCF (Groupe Hospitalier Pitié-Salpêtrière Charles Foix) neurology department 2 for a diagnosis of low grade glioma or anaplastic glioma with loss 1p / 19q sub-reserve histo-molecular confirmation after national reading (POLA) and presenting:

   * An MSISQ15 (Multiple Sclerosis Intimacy and Sexuality Questionnaire) questionnaire with at least one of the items rated "4" or "5" and
   * A HAD (Hospital Anxiety and Depression) questionnaire (depression component) with a score ≤ 11
2. Any major patient with MS(Multiple Sclerosis), followed in the GHPSCF Department of Neurology:

   * With an EDSS (Expanded Disability Status Scale) greater than or equal to 1 and
   * An MSISQ15 questionnaire with at least one of the items rated "4" or "5".
   * A HAD questionnaire (depression component) with a score ≤ 11
3. Signature of informed consent
4. Patient affiliated to a social security system

Exclusion Criteria:

1. Minor patients
2. Pregnant women
3. Patients who do not understand and / or speak French and / or are unable to sign consent
4. Patients with neurological impairment
5. Patients with chronic sexual disorders who have already received treatment.
6. Patients with a HAD score (depression component) greater than 11
7. Patients with MS who had a corticosteroid-treated outbreak in the last two months.
8. Patients with low-grade glioma with clinical and / or radiological scalability during the last three months
9. Any patient whose alteration of the general state would not allow to follow the program.
10. Patients under legal protection

For patient's partners:

Inclusion criteria:

1. Any patient partner, whose patient has wished to participate and who has accepted.
2. Signing of informed consent

Non-Inclusion Criteria:

1. Minor partners
2. Pregnant women
3. Any person who does not understand and / or speak French and / or is unable to sign the consent
4. Partners under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-07-26 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-07-26 (Estimated)

PRIMARY OUTCOMES:
Change of MSISQ15 (Multiple Sclerosis Intimacy and Sexuality Questionnaire) | Inclusion and 3 months
  Change of MSISQ15 sexual dysfunctional items at 3-months from baseline

SECONDARY OUTCOMES:
Change of MSISQ15 (Multiple Sclerosis Intimacy and Sexuality Questionnaire) | Inclusion and 6-months
  Change of MSISQ15 sexual dysfunctional items at 6-months from baseline
Change of HAD scale (Hospital Anxiety and Depression) | Inclusion and 3 months
  Change of HAD scale score at 3-months from baseline
Change of HAD scale (Hospital Anxiety and Depression) | Inclusion and 6 months
  Change of HAD scale score at 6-months from baseline
Change of Rosenberg's Self-esteem Scale | Inclusion and 3 months
  Change of Rosenberg's Self-esteem Scale score at 3-months from baseline
Change of Rosenberg's Self-esteem Scale | Inclusion and 6 months
  Change of Rosenberg's Self-esteem Scale score at 6-months from baseline
Change of Quality of life scale | Inclusion and 3 months
  Change of Quality of life scale score at 3-months from baseline
Change of Quality of life scale | Inclusion and 6 months
  Change of Quality of life scale score at 6-months from baseline
Change of QLQ-C30/BM20 scale (Quality of Life Questionnaire - Core Questionnaire / Brain Module) | Inclusion and 3 months
  Change of QLQC30/BM20 score at 3-months from baseline
Change of QLQ-C30/BM20 scale (Quality of Life Questionnaire - Core Questionnaire / Brain Module) | Inclusion and 6 months
  Assessment of QLQC30/BM20 score at 6-months from baseline
Change of SEP59 scale (Sclérose En Plaques) | Inclusion and 3 months
  Change of SEP59 scale score at 3-months from baseline
Change of SEP59 scale (Sclérose En Plaques) | Inclusion and 6 months
  Change of SEP59 scale score at 6-months from baseline
Program satisfaction scale | 3 months
  Program satisfaction scale scores at 3-months
Program satisfaction scale | 6 months
  Program satisfaction scale scores at 6-months

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Pitie Salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: No